CLINICAL TRIAL: NCT02220595
Title: A Comparison of Cognitive Function After Carotid Endarterectomy and Stenting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Panos Kougias, Chief, Vascular Surgery, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H - 22797
Record Dates: First submitted 2014-08-08; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Carotid Artery Occlusive Disease
Keywords: Stenting; Endarterectomy; Cognition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carotid stenting (Experimental): Carotid artery stenting for treatment of carotid artery stenosis
  Interventions: Procedure: Carotid endarterectomy vs. carotid stenting
- Carotid endarterectomy (Active Comparator): Carotid artery endarterectomy for treatment of carotid artery stenosis
  Interventions: Procedure: Carotid endarterectomy vs. carotid stenting

INTERVENTIONS:
Procedure: Carotid endarterectomy vs. carotid stenting

SUMMARY:
This study compares cognitive function after carotid endarterectomy and stenting.

ELIGIBILITY:
Inclusion Criteria:

* Carotid artery occlusive disease, asymptomatic greater than 80% with CTA or carotid duplex

Exclusion Criteria:

* Contraindication for carotid endarterectomy or stenting

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Difference in RAVLT score | Six weeks

SECONDARY OUTCOMES:
Cognitive tests for attention, memory, processing speed, mood, motor function, visual-spatial skills, executive functioning | Six weeks and six months
Cognitive tests of attention | Six weeks
  Comparison in cognitive tests for attention between carotid endarterectomy and stenting
Cognitive tests for memory | Six weeks
  Comparison in cognitive tests for memory between carotid endarterectomy and stenting
Cognitive tests for processing speed | Six weeks
  Comparison in cognitive tests for processing speed between carotid endarterectomy and stenting
Cognitive tests of mood | Six weeks
  Comparison in cognitive tests for mood between carotid endarterectomy and stenting
Tests of motor function | Six weeks
  Comparison in cognitive tests for motor function between carotid endarterectomy and stenting
Cognitive tests of visual-spatial skills | Six weeks
  Comparison in cognitive tests of visual-spatial skills between carotid endarterectomy and stenting
Cognitive tests of executive functioning | Six weeks
  Comparison in cognitive tests for executive functioning between carotid endarterectomy and stenting
Cognitive tests of attention | Six months
  Comparison in cognitive tests for attention between carotid endarterectomy and stenting
Cognitive tests of memory | Six weeks
  Comparison in cognitive tests for memory between carotid endarterectomy and stenting
Cognitive tests of processing speed | Six months
  Comparison in cognitive tests for processing speed between carotid endarterectomy and stenting
Cognitive tests of mood | Six months
  Comparison in cognitive tests for mood between carotid endarterectomy and stenting
Tests of motor function | Six months
  Comparison in cognitive tests for motor function between carotid endarterectomy and stenting
Cognitive tests of visual-spatial skills | Six months
  Comparison in cognitive tests for visual-spatial skills between carotid endarterectomy and stenting
Cognitive tests of executive functioning | Six months
  Comparison in cognitive tests for executive functioning between carotid endarterectomy and stenting
Difference in new ischemic infarcts in Diffusion - weighted MRI | Six weeks
  Difference in new ischemic infarcts in Diffusion - weighted MRI
Difference in new ischemic infarcts in Diffusion - weighted MRI | Six months
  Difference in new ischemic infarcts in Diffusion - weighted MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Michael E. Debakey VAMC, Houston, Texas, United States